CLINICAL TRIAL: NCT06937515
Title: EVALUATION OF THE EFFICACY OF AN ANTIMELANOGENESIS AGENT (MELASYL) IN DIFFERENT CONCENTRATIONS UNDER PART OF VISIBLE LIGHT [400-450NM] EXPOSURES AND UNDER FULL VISIBLE LIGHT [400-700NM] EXPOSURES
Brief Title: MELASYL EFFICACY UNDER PART OF VISIBLE LIGHT
Acronym: BIOVI2
Status: Completed | Type: Observational
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Other Study IDs: ACR_BIOVI2_23-02381
Record Dates: First submitted 2025-04-20; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Visible Light Exposure on Healthy Back Skin
Keywords: pigmentation; visible light; full visible light

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Melasyl at 1% and 0.5% versus its vehicle under High Energy Visible light or full visible light: A total of eight (8) zones of 3x3cm will be delineated on the back, four (4) zones per hemi-back (left and right) and exposed under UVA1+physical multilayer filter cut-off wavelengths under 400nm for [400-450nm] OR exposed under full visible light for [400-700nm].
  - Three (3) zones per hemi-back will be treated with topical treatments during the 7 weeks of the study: IP1: Melasyl 1% in Bright Matte (893286 03) IP2: Melasyl 0.5% in Bright Matte (893286 02) IP3: Bright Matte vehicle (893286 P)
  - One (1) zone per hemi-back will not be treated (control NT)
  Interventions: Other: Cosmetic topical products

INTERVENTIONS:
Other: Cosmetic topical products — Cosmetic topical products efficacy evaluation

SUMMARY:
The study intends to evaluate the efficacy of an anti-melanogenesis active in different concentrations under part of visible Light [400-450nm] exposures and under full visible light [400-700nm] exposures.

It is carried out on cosmetic products for which the safety has been assured by a toxicologist, with the aim of confirming the efficacy of the products, which will be used by a large number of consumers under normal and reasonably foreseeable use conditions.

DETAILED DESCRIPTION:
The main objective of this study is to assess the efficacy of an anti-melanogenesis active in different concentrations under [400-450nm] exposures and under [400-700nm] in healthy volunteers by skin colorimetry (Delta E).

The secondary objectives are:

* To assess the efficacy of anti-melanogenesis active in different concentrations under [400-450nm] exposures and under [400-700nm] exposures in healthy volunteers by clinical evaluation and additional colorimetry measurements (Delta L*, a*, b* and ITA°).
* To assess the local tolerance and safety of the topical formulations under [400-450nm] exposure and under [400-700nm] by recording adverse events and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female or male volunteer from 18 to 65 years old
2. Skin type III-IV according to the Fitzpatrick classification
3. Average ITA° (Individual Typologic Angle calculated value) on the back between 18° and 34° at screening and inclusion visits with an allowed difference of ± 2° between screening and inclusion visits
4. Uniform skin color over the eight zones (difference in ITA° between each zone should not be more than 4°)
5. Absence of freckles, naevi, hypo or hyper pigmented regions, hairs and marks of bronzing on the investigational area on the back
6. Female subject of childbearing potential, who is not sexually active, or using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study or menopausal female (with absence of menstruations for less than one year) or post-menopausal female (with absence of menstruations for more than one year)
7. Female of childbearing potential or menopausal female (with absence of menstruations for less than one year) willing to undergo urine pregnancy test
8. Subject willing and able to fulfil the study requirements and schedule
9. Subject informed about the study objectives and procedures, and able to understand them
10. Subject who has given written inform consent

Exclusion Criteria:

1. Subject who is pregnant or lactating or who is planning to become pregnant during the study
2. Subject with BMI > 30
3. Having planned UV exposure of the investigational area (sunlight or sunbeds) throughout the study
4. Having used sunbeds or had excessive sun exposure of the investigational area within the 3 months before inclusion
5. Having sunburn (erythema) on the back
6. Dermatological disorders affecting the investigational area (presence of naevi, freckles, excess hair or uneven skin tones, vitiligo, photo-dermatological problems
7. History of skin cancer
8. History of abnormal response to sun
9. Presence of recent suntan (according to Investigator opinion) or photo-test marks
10. History of allergy, hypersensitivity, or any serious reaction to any cosmetic product
11. Any concomitant medical condition that may interfere with the study conduct in the opinion of the investigator
12. Having used within the month before inclusion any systemic medication for more than 5 consecutive days (e.g. steroidal and non-steroidal anti-inflammatory drugs, corticoids, insulin, antihistamines, antihypertensive, antibiotics such as quinolone, tetracycline, thiazides, fluoroquinolones)
13. Having used within the month before inclusion any medication known to cause abnormal responses to UV exposure (e.g. vitamin A derivative, psoralen, aminolevulinic acid derivatives, etc.), or having planned to use these medications during the study
14. Having used within the 3 months before inclusion any depigmenting / whitening or pro-pigmenting topical treatments, or any systemic treatment that would interfere with the study assessments (anti-inflammatory drugs, corticoids, retinoids, hydroquinone, etc.) or having planned to use these treatments during the study
15. Having used, within the past 6 months, any physical treatment including laser or phototherapy (PUVA, IPL, PDT…) on the investigational area, or having planned to use these treatments during the study
16. Having planned to perform intensive sport (> 5 hours per week) or swim during the study
17. Subject who declares to be deprived of freedom by administrative or legal decision
18. Subject who cannot be contacted by telephone in case of emergency
19. Subject having participated within the 30 days before inclusion or currently participating in another clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female volunteers from 18 to 65 yo, with Fitzpatrick III and IV and an ITA° between 18° to 34° at screening.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Skin color measurement | from Day 1 to Day 47.
  Measurement of the skin color using Chromameter® (non-invasive assessment) between the exposed zone (ZE) and non-exposed zone (ZNE).

SECONDARY OUTCOMES:
Visual scoring of pigmentation | from Day 1 to Day 47.
  Visual evaluation of the pigmentation using L'Oreal pigmentation scale (0-13 points)
Visual scoring of erythema | from Day 1 to Day 47.
  Visual evaluation of the erythema using L'Oreal pigmentation scale (0-13 points)

OTHER OUTCOMES:
Safety assessment | from Day 1 to Day 47.
  Safety will be assessed by recording Adverse Events, including cutaneous reactions (local intolerance), from the informed consent form signature date until the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Romania, Budapest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piffaut V, De Dormael R, Belaidi JP, Bertrand L, Passeron T, Bernerd F, Marionnet C. Topical prevention from high energy visible light-induced pigmentation by 2-mercaptonicotinoyl glycine, but not by ascorbic acid antioxidant: 2 randomized controlled trials. Front Pharmacol. 2025 Oct 9;16:1651068. doi: 10.3389/fphar.2025.1651068. eCollection 2025. PMID 41142247